CLINICAL TRIAL: NCT04417439
Title: Turgut Özal Medical Center
Brief Title: The Effect of Acute Phase Treatment Approaches on Creatine Kinase and the Musculoskeletal System in Different Types of Burns
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Engin Ramazanoglu, Principal Investigator, Inonu University
Other Study IDs: ERamazanoglu
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Burn Injury
Keywords: Acute-phase burn; Creatine Kinase, MM Form,; Musculoskeletal Development; Treatment Effectiveness
MeSH Terms: conditions — Burns | interventions — Creatine Kinase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- flame burns: The joint range of motion was assessed by a universal goniometer within the affected areas of burn patients. A tape measure with a width of 7 mm was used to evaluate the circumference measurement in individuals. The biochemical examination of CK (creatine kinase) was performed in the laboratories.
  Interventions: Other: universal goniometer. evaluate the circumference measurement. The biochemical examination of CK (creatine kinase)
- scald burns: The joint range of motion was assessed by a universal goniometer within the affected areas of burn patients. A tape measure with a width of 7 mm was used to evaluate the circumference measurement in individuals. The biochemical examination of CK (creatine kinase) was performed in the laboratories.
  Interventions: Other: universal goniometer. evaluate the circumference measurement. The biochemical examination of CK (creatine kinase)
- electrical burns: The joint range of motion was assessed by a universal goniometer within the affected areas of burn patients. A tape measure with a width of 7 mm was used to evaluate the circumference measurement in individuals. The biochemical examination of CK (creatine kinase) was performed in the laboratories.
  Interventions: Other: universal goniometer. evaluate the circumference measurement. The biochemical examination of CK (creatine kinase)

INTERVENTIONS:
Other: universal goniometer. evaluate the circumference measurement. The biochemical examination of CK (creatine kinase) — The joint range of motion within the affected areas of burn patients was assessed by a universal goniometer. A 7-mm-wide tape measure was used to evaluate circumference measurement in individuals. The biochemical analysis of CK (creatine kinase) was performed by an expert on blood samples taken from patients in the hospital laboratories.

SUMMARY:
There are very few studies indicating the effect of acute phase treatment approaches on creatine kinase and the musculoskeletal system in the physiotherapy and rehabilitation process. Rehabilitation in burn patients is a benchmark due to return to pre-burn life. Therefore, this study was conducted to determine the effect of acute phase treatment approaches on creatine kinase and the musculoskeletal system in different types of burns.

DETAILED DESCRIPTION:
In the literature, there are very few objective and quantitative studies comparing the effects of standard wound care and rehabilitation period on different burn types in burn patients. Thus, our study was designed to investigate the effects of acute phase treatment approaches on creatine kinase and the musculoskeletal system in different types of burns.

ELIGIBILITY:
Inclusion Criteria:

* the study were being aged between 18-65 years and having different burn types, and flame, scald, and electrical burns were included in the study.
* The burn percentage and mortality percentage were calculated, and patients with a burn percentage of less than fifty percent were included.

Exclusion Criteria:

* the study were having a systemic disease, having substance abuse, and having a burn percentage of more than fifty percent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 37 individuals, including 10 females and 27 males
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-05-12 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
universal goniometer | three weeks
  Universal goniometer was used to measure arm flexion movement.
A tape measure with a width of 7 mm | three weeks
  Anthropometric measurement (arm circumference measurement) was made with a tape measure of 7 mm width.
The biochemical examination of CK (creatine kinase) | three weeks
  Creatine kinase concentration in the blood was evaluated.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Malatya İnönü University, Malatya
  - Turgut Özal medical center, Malatya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flores O, Tyack Z, Stockton K, Ware R, Paratz JD. Exercise training for improving outcomes post-burns: a systematic review and meta-analysis. Clin Rehabil. 2018 Jun;32(6):734-746. doi: 10.1177/0269215517751586. Epub 2018 Jan 10. PMID 29320878
- [Background] Goverman J, Mathews K, Goldstein R, Holavanahalli R, Kowalske K, Esselman P, Gibran N, Suman O, Herndon D, Ryan CM, Schneider JC. Adult Contractures in Burn Injury: A Burn Model System National Database Study. J Burn Care Res. 2017 Jan/Feb;38(1):e328-e336. doi: 10.1097/BCR.0000000000000380. PMID 27380122